CLINICAL TRIAL: NCT06091046
Title: Assessment of Discomfort in Intensive Care Patients and Psychometric Testing of the Applied Questionnaire IPREA-N
Brief Title: Discomfort in Intensive Care Patients - IPREA-N
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); The Hospital of Vestfold (Other); Ostfold Hospital Trust (Other); Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Helene Berntzen, RN, CCN, Phd, Oslo University Hospital
Other Study IDs: 612620
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Discomfort
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate discomforts experienced by intensive care patients during their critical illness period. We will use the Norwegian version of the questionnaire Inconforts des Patients de REAnimation (IPREA), the IPREA-N.Patients will be asked to rate18 questions about different possible discomforts on a 0-10 scale after their intensive care stay. Furthermore we aim to test whether the questionnaire when translated into Norwegian is useful in the Norwegian patient population.

The aim of the study is

* to assess perceived discomfort in intensive care patients using the IPREA-N questionnaire
* to test psychometric properties of the questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients (> 18 years),
* Understanding Norwegian
* Having spent more than 48 hours in the intensive care unit.
* Ability to consent to participation and self-report discomfort

Exclusion Criteria:

* Patients who move to another hospital and cannot complete the questionnaire within 24 hours due to health status or practical reasons.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intensive care units at five different hospitals in the South-East Norway will participate in the study. Each hospital will include approximately 50 patients.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Discomfort measured by IPREA-N questionnaire | Within 24 hours following Intensive care unit stay
  IPREA-N consists of 18 Questions about discomfort during intensive care stay, answered on a 0-10 scale. Questions cover discomforts caused by noise, too much light, uncomfortable bed, lack of sleep, thirst, hunger, feeling cold, feeling hot, pain, medical devices, embarrassment, anxiety or panic, isolation, visiting hours restriction, lack of telephone, lack of information, difficulty breathing and feelings of depression,

CONTACTS AND LOCATIONS:
Overall Officials: Helene Berntzen, Phd, Principal Investigator — Oslo University Hospital